CLINICAL TRIAL: NCT04731181
Title: Mobile App (Little Lovely Dentist) Versus Tell-Show-Do Technique in Reduction of Anxiety and Pain During Administration of Local Anaesthesia in Children (A Randomized Clinical Trial)
Brief Title: Effectiveness of Mobile Applications During the Administration of Local Anesthesia in Pediatric Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marian Mamdouh Sedky Reda, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: mobile app in dentistry
Record Dates: First submitted 2021-01-19; First posted 2021-01-29 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: parallel-group and allocation ratio (1:1) Intervention: mobile application (little lovely dentist). Control: Tell-Show-Do technique.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile application (little lovely dentist). (Experimental): intervention mobile application simulating the dental procedure that will be done to the child
  Interventions: Behavioral: mobile application (little lovely dentist).
- Tell-Show-Do technique. (No Intervention): control behavior technique where ''tell'' is to tell the child about the procedure in non-threatening words, ''show'' is to demonstrate the procedure to the child, and ''do'' is the execution of the procedure

INTERVENTIONS:
Behavioral: mobile application (little lovely dentist). — mobile application
  Arms: mobile application (little lovely dentist).

SUMMARY:
To evaluate the mobile games' effect on patient acceptance of local anesthesia and decreasing dental pain and anxiety levels in pediatric patients.

DETAILED DESCRIPTION:
a randomized clinical trial with parallel-group and allocation ratio (1:1). intervention group: mobile application (little lovely dentist) control group: Tell-Show-Do technique. in children aged 4-6 years who need local anesthesia for dental treatment during their first dental visit.

For both groups:

Verbal assent from participating patients and written consent from their legal guardians will be taken.

1. Taking personal data, medical and dental history.
2. Diagnosis and determination of the required treatment.
3. Measuring preoperative anxiety using a pulse oximeter.
4. Evaluate preoperative anxiety using RMS-pictorial scale.
5. Using the behavior guidance technique:

   Intervention group: Allow the child to play the module simulating the required procedure. Control group: tell-show-do technique is used to explain the procedure to the child
6. Administration of local anesthesia and evaluation of child behaviour during the administration of local anaesthesia using Venham's behaviour rating scale and Frankl behaviour rating scale .
7. Measuring postoperative anxiety using the pulse oximeter.
8. Evaluate postoperative anxiety using RMS-pictorial scale.
9. Evaluate postoperative pain using the visual analog scale.

in second visit (after 1 week)

1) Evaluation of child behavior during the second dental visit using Venham's behavior rating scale and Frankl behavior rating scale. outcome:

1. ry: Pre and postoperative anxiety using Pulse oximeter and RMS-pictorial scale.
2. ry: Postoperative pain using Visual analog scale, evaluation of attitude during the administration of local anaesthesia at first and second dental visits using -Venham's behavior rating scale-Frankl behavior rating scale. the study will be held in 2 visits.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-6 years.
* Children without any systemic or mental disorders.
* Children without any prior experience with the dental environment or treatment procedures (first dental visit).
* Children whose behavior could be rated as positive or negative based on the Frankl behavior rating scale.

Exclusion Criteria:

* Children seeking dental treatment that does not necessitate local anesthesia.
* Children suffering from any systemic or mental disorders.
* Children who are not willing to participate in the study

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | before administration of local anesthesia during the first dental visit
  Preoperative anxiety will be measured before administration of local anesthesia using a fingertip pulse oximeter (IMDK) in beat per minute unit (BPM)
postoperative anxiety | immediately after administration of local anesthesia during the first dental visit
  postoperative anxiety will be measured immediately after administration of local anesthesia using a fingertip pulse oximeter (IMDK) in beat per minute unit (BPM)
Preoperative anxiety score | before administration of local anesthesia during the first dental visit
  will be assessed by RMS-pictorial scale ( Raghavendra, Madhuri, Sujata - pictorial scale) before administration of local anesthesia in a numerical unit from 1-5 where 1 denotes the minimum anxiety and 5 denotes the maximum anxiety
post-operative anxiety score | immediately after administration of local anesthesia during the first dental visit
  will be assessed by RMS-pictorial scale ( Raghavendra, Madhuri, Sujata - pictorial scale) immediately after administration of local anesthesia in a numerical unit from 1-5 where 1 denotes the minimum anxiety and 5 denotes the maximum anxiety

SECONDARY OUTCOMES:
Postoperative pain | immediately after administration of local anesthesia during the first dental visit
  Postoperative pain will be measured immediately after administration of local anesthesia by the visual analog scale in a numerical unit 0-10 where 0 denotes no pain and 10 denotes the worst pain
Attitude during the first and second dental visits using frankle behavior rating scale | during administration of local anasthesia during the the first and second dental visits (after 1 week)
  evaluation of child behavior during the first and second visits using frankle behavior rating scale in a numerical unit rating 1-4 where,
  1. Definitely Negative:
     Refusal of treatment, crying forcefully, fearful, or any other overt evidence of extreme negativism.
  2. Negative:
     Reluctant to accept treatment, uncooperative, some evidence of negative attitude but not pronounced withdrawn.
  3. Positive:
     Acceptance of treatment; at times curious, willing to comply with the dentist, at times with reservation but patient follows the dentist's directions cooperatively
  4. Definitely positive:
  Good rapport with the dentist, interested in dental procedures, and laughing and enjoying the situation.
Attitude during the first and second dental visits using Venham's behavior rating scale | during administration of local anasthesia during the first and second dental visits (after 1 week)
  evaluation of child behavior during the first and second visits using Venham's behavior rating scale in a numerical unit using score 0-3 where, 0- Total cooperation, best working conditions, no crying, or physical protest.
  1. Mild, soft verbal protest or quiet crying as a signal of discomfort, but doesn't obstruct progress. Appropriate behavior for the procedure.
  2. Protest more prominent. Both crying and hand signals. May move head around making it hard to perform the treatment. Protest more distracting and troublesome. However, the child still complies with the request to cooperate.
  3. Protest presents a real problem to the dentist. Complies with demands reluctantly, requiring more effort by dentist + Body movement.

CONTACTS AND LOCATIONS:
Overall Officials: Passant Nagi, PHD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

REFERENCES:
- [Result] Steimer T. The biology of fear- and anxiety-related behaviors. Dialogues Clin Neurosci. 2002 Sep;4(3):231-49. doi: 10.31887/DCNS.2002.4.3/tsteimer. PMID 22033741
- [Result] Saatchi M, Abtahi M, Mohammadi G, Mirdamadi M, Binandeh ES. The prevalence of dental anxiety and fear in patients referred to Isfahan Dental School, Iran. Dent Res J (Isfahan). 2015 May-Jun;12(3):248-53. PMID 26005465
- [Result] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259
- [Result] Ghanei M, Arnrup K, Robertson A. Procedural pain in routine dental care for children: a part of the Swedish BITA study. Eur Arch Paediatr Dent. 2018 Oct;19(5):365-372. doi: 10.1007/s40368-018-0368-2. Epub 2018 Sep 7. PMID 30194611
- [Result] Shetty RM, Khandelwal M, Rath S. RMS Pictorial Scale (RMS-PS): an innovative scale for the assessment of child's dental anxiety. J Indian Soc Pedod Prev Dent. 2015 Jan-Mar;33(1):48-52. doi: 10.4103/0970-4388.149006. PMID 25572374
- [Result] Monteiro J, Tanday A, Ashley PF, Parekh S, Alamri H. Interventions for increasing acceptance of local anaesthetic in children and adolescents having dental treatment. Cochrane Database Syst Rev. 2020 Feb 27;2(2):CD011024. doi: 10.1002/14651858.CD011024.pub2. PMID 32104910
- [Result] Saxena P, Gupta SK, Newaskar V, Chandra A. Advances in dental local anesthesia techniques and devices: An update. Natl J Maxillofac Surg. 2013 Jan;4(1):19-24. doi: 10.4103/0975-5950.117873. PMID 24163548
- [Result] Behavior Guidance for the Pediatric Dental Patient. Pediatr Dent. 2017 Sep 15;39(6):246-259. No abstract available. PMID 29179365
- [Result] Radhakrishna S, Srinivasan I, Setty JV, D R MK, Melwani A, Hegde KM. Comparison of three behavior modification techniques for management of anxious children aged 4-8 years. J Dent Anesth Pain Med. 2019 Feb;19(1):29-36. doi: 10.17245/jdapm.2019.19.1.29. Epub 2019 Feb 28. PMID 30859131